CLINICAL TRIAL: NCT06324214
Title: Urolithin A Supplementation During Pulmonary Rehabilitation Participation in Patients With Chronic Obstructive Pulmonary Disease: a Randomized Pilot and Feasibility Study
Brief Title: Oral Supplementation During PR Participation in COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Amazentis SA (Industry)
Responsible Party: Principal Investigator, Bryan Ross, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-9352
Record Dates: First submitted 2024-03-04; First posted 2024-03-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants will participate in a standard PR program and will receive placebo.
  Interventions: Other: Placebo
- Intervention (Urolithin A: Mitopure) Group (Active Comparator): Participants will participate in a standard PR program and will receive the oral supplement.
  Interventions: Dietary Supplement: Urolithin A (Mitopure)

INTERVENTIONS:
Dietary Supplement: Urolithin A (Mitopure) — Compound belonging to the 'urolithin' class. First discovered over 40 years ago as a gut-derived metabolite in rats and subsequently in humans. A food and dietary ingredient, and more specifically, a post-biotic compound. Derived from ellagitannins, which are present in foods such as pomegranate, berries, and walnuts. An 'inducer' of mitophagy.
  Arms: Intervention (Urolithin A: Mitopure) Group
Other: Placebo — Placebo.
  Arms: Placebo Group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a very common and chronic lung condition and is a leading cause of morbidity and death. These patients have persistent breathlessness and exercise intolerance, affecting their ability to carry out routine daily tasks. Standard COPD treatments include medicines/puffers as well as participation in a Pulmonary Rehabilitation (PR) program. PR programs are delivered by a diverse team of healthcare experts in exercise and nutrition. It is possible that an emerging nutritional oral supplement could target the muscular dysfunction seen in patients with COPD in part by promoting better working mitochondria, the energy 'engine' of muscle. A series of recently published studies in sedentary adults and in older adults have demonstrated the safety, tolerability, and potential clinical effectiveness of this supplement.

In this regard, the investigators plan to lead a large randomized controlled trial (RCT) to test whether oral supplementation in patients with COPD who are also participating in a standard PR program will improve overall exercise performance. The investigators will also test muscle strength, cognition, body composition, and other clinically important outcomes such as quality of life. Lastly, the investigators will use muscle tissue from a subgroup of volunteers to investigate the effect on muscle/mitochondrial structure/function.

The focus is actually the critical 'first step' before the larger RCT: a pilot and feasibility study on a smaller number of participants with COPD, as an important proof-of-concept that the larger study can, and should, be conducted.

DETAILED DESCRIPTION:
The main objectives for this pilot feasibility study are to document recruitment rates, collect information on participant acceptability of tests, establish the capacity to run the RCT at our site, to demonstrate successful molecular testing of specimens, and to generate pilot data for the outcomes being tested in the larger subsequent RCT.

The overarching goal for the 'larger', future project will be to determine the effect of the oral supplement on exercise capacity, muscle strength, mitochondrial function, health-related quality of life, cognition, symptom burden, and safety/adherence in patients with COPD who are participating in a Pulmonary Rehabilitation program. The goal of the present research project is to complete a pilot and feasibility study testing the same clinical outcomes on a smaller sample of eligible study participants during which participants receive the intervention for 8 weeks.

The primary objective is to determine whether administration of the oral supplement during participation in a standard multi-week in-person Pulmonary Rehabilitation (PR) program is associated with an improvement in exercise endurance capacity in patients with COPD, compared with PR participation and placebo supplementation.

The secondary objectives are to determine the effect of the oral supplement on i) global conditioning and exercise capacity; ii) muscle strength; iii) mitochondrial function; iv) body composition; v) quality of life and burden of disease; vi) cognition; vii) adverse events/complications and adherence, and viii) blood levels of Urolithin A.

We hypothesize that patients with COPD receiving oral supplementation during PR participation will demonstrate an improvement in Constant Work Rate Exercise Test (CRWET) time after 8 weeks when compared to patients with COPD who receive placebo and PR participation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, aged >40, former smokers with ≥10 pack-year smoking history
2. Post-bronchodilator forced expiratory volume at one second (FEV1) / forced vital capacity (FVC) ratio < 0.7, with FEV1 < 80% (moderate, Global Initiative for Chronic Obstructive Lung Disease '(GOLD) 2') FEV1 < 50% (severe, 'GOLD 3') or FEV1 < 30% (very severe, 'GOLD 4') COPD
3. Baseline 6MWD of ≥50m
4. Prior receipt of at least 2 doses of the Coronavirus Disease of 2019 (COVID-19) vaccine

Exclusion Criteria:

1. Inability to participate in a standard PR program
2. Severe/unstable cardiac disease, neurological or orthopedic conditions which could hinder exercise performance
3. Inability to provide consent due to language or cognitive barrier
4. Previous PR participation in the last 12 months, or in a study involving an exercise program in the last 6 months
5. Experienced an exacerbation of COPD (ECOPD) within the prior 4 weeks
6. Long-term oxygen therapy use, or maintenance oral corticosteroid use
7. Presence of pacemaker or implantable cardioverter defibrillator (ICD) (unless participant opts out of bioelectrical impedance assay)
8. Unwilling to agree to refrain from using, or are found to be using, the following supplementary antioxidant vitamins from 7 days prior to dosing and throughout the treatment period: Coenzyme Q10, resveratrol, and L-carnitine
9. Unwilling to agree to refrain from using, or are found to be using, the following dietary restrictions from 7 days prior to dosing and throughout the treatment period: pomegranate juice, walnuts, pecans, strawberries, raspberries, and blackberries
10. Allergy to lecithin, to soy or to sunflower
11. Pregnant, breastfeeding or planning to become pregnant
12. Use of anticoagulant or presence of a clotting disorder (if participating in muscle biopsy subgroup)
13. Allergy to anesthetics such as xylocaine and lidocaine (if participating in muscle biopsy subgroup)
14. Chronic myalgia, fibromyalgia or conditions characterized by regular muscle pain (if participating in muscle biopsy subgroup)
15. Metal fixation plates or screws in the legs from a previous surgery (if participating in muscle biopsy subgroup)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Constant Work Rate Exercise Test (CRWET) | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Exercise test whereby the workload is constant and is calculated as a percentage of the peak power output observed in the incremental test.

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  6-Minute Walk Distance (6MWD) obtained on a standard 6MWT
Quadriceps strength | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  4-second maximum quadriceps strength test
Mitochondrial function | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Fresh samples
Muscle histology | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Stains for mitochondrial markers (including succinate dehydrogenase (SDH)): post-intervention in comparison to pre-intervention.
Tissue microscopy | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Transmission electron microscopy for assessment of number of mitochondria: post-intervention in comparison to pre-intervention.
Tissue microscopy | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Transmission electron microscopy for assessment of morphology of mitochondria: post-intervention in comparison to pre-intervention.
Specific protein detection | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Targeted Western blot analysis for proteins related to mitochondrial function: post-intervention in comparison to pre-intervention.
RNA analyses | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Specific mRNA transcript changes related to mitochondrial function and whole transcriptome changes: post-intervention in comparison to pre-intervention.
Body composition | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Dual X-ray absorptiometry (DXA) scan
Body impedance | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Bioelectrical impedance assay (BIA)
Disease-specific impact on quality of life | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  St. George's respiratory questionnaire (SGRQ)
Burden of disease | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  COPD assessment test (CAT)
Cognition | Pre-intervention (baseline) and Post-intervention (after 8 weeks)
  Stroop test
Adverse events | 12 weeks
  Adverse events (AEs) will be monitored from the signing of the Informed Consent Form (ICF) through completion of study participation. If any AEs do occur, study participants will be followed until symptoms have resolved or have returned to baseline levels. All outstanding AEs will be followed until resolution or until the participant's last study visit.
Differences in dosed missed | 8 weeks
  The total number of doses missed will be recorded and reported.
Blood levels of the intervention | Day 28
  Blood levels of Urolithin A will be collected at the mid-point of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No